CLINICAL TRIAL: NCT05768815
Title: Optimizing Mental Health for Infants Exposed to Early Adversity: A Comparative Effectiveness Trial of the Breaking the Cycle and Maxxine Wright Intervention Programs
Brief Title: Optimizing Mental Health for Infants Exposed to Early Adversity: A Comparison of Breaking the Cycle and Maxxine Wright
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-02-23-8940
Record Dates: First submitted 2023-02-23; First posted 2023-03-14 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-03

CONDITIONS: Mother-Child Relations; Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breaking the Cycle Intervention group (Experimental)
  Interventions: Behavioral: Breaking the Cycle Program
- Maxxine Wright Intervention group (Active Comparator)
  Interventions: Behavioral: Maxxine Wright Program

INTERVENTIONS:
Behavioral: Breaking the Cycle Program — BTC is a prevention and early intervention program in Toronto, Canada, serving substance-using pregnant and/or parenting women with children under six years of age. Established by the Canadian Mothercraft Society in 1995, BTC is funded by the Community Action Program for Children and the Canadian Prenatal Nutrition Program through the Public Health Agency of Canada. BTC provides three program components that act synergistically: a) individualized services for mothers, b) individualized services for children, and c) relational interventions that enhance the mother-child relationship and promote infant mental health. Coordinated supports are offered through formal partnerships across service sectors. In 2004, BTC was recognized by the United Nations as an exemplary program serving pregnant and parenting women with substance use problems, and their young children.
  Arms: Breaking the Cycle Intervention group
Behavioral: Maxxine Wright Program — Founded in 2005 and located in Surrey, British Columbia, the Maxxine Wright Community Health Centre (MWCHC) supports women who are pregnant and/or have young children and are impacted by substance use and/or violence. Women do not need to have children in their care to receive services. The program is funded and operated by the Fraser Health Authority, with additional in-kind support from the BC Ministry for Children and Family Development and the BC Ministry of Social Development and Poverty Reduction. MW addresses maternal substance use and exposure to violence through women-centered, trauma-informed, culturally grounded, and interdisciplinary approaches. Primary services offered include addiction counselling, primary health care, and group therapy to address interpersonal violence. Within MW, child-focused services are limited to primary health (e.g., well baby checks, childcare).
  Arms: Maxxine Wright Intervention group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of the Breaking the Cycle (BTC) and Maxxine Wright (MW) programs in substance-involved mothers and their children. One key difference between the two programs is that the BTC program contains an infant mental health component while the MW program primarily focuses on the mothers. The main questions the trial aims to answer are:

* Do children at BTC demonstrate enhanced infant mental health compared to children at MW up to 2 years post-intervention?
* Do mother-child dyads at BTC experience more decreases in child adverse childhood experiences (ACE), maternal stress, and mental health symptoms and have better home environment scores, parenting attitudes, and mother-child relationship scores compared to mother-child dyads at MW?
* Are enhanced infant mental health outcomes associated with children's lower psychosocial risk scores and mothers with lower ACE scores, lower depression and anxiety scores, and lower maternal stress?
* Are the associations between treatment dose and infant mental health scores mediated by parenting attitudes and the mother-child relationship? Does child exposure to psychosocial risk moderate the association between treatment dose and child outcomes?
* How do the mechanisms of change lead to the effectiveness of BTC? What are the potential lifetime health and non-health outcomes of at-risk children at BTC? What is the long-term social return on investment (SROI) of BTC?

Participants will complete several questionnaires at three timepoints while receiving services at either BTC or MW: during the intake phase, 12 months after their engagement in services and 24 months after their engagement in services.

Given that the two programs serve a similar demographic of women, researchers will compare the BTC group and the MW group to establish the comparative effectiveness and mechanisms of change of the infant mental health component of BTC.

ELIGIBILITY:
Inclusion Criteria:

* receiving services at either BTC or MW
* having a child under the age of 6 years
* being able to answer a questionnaire in English

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Children's socio-emotional functioning will be measured using the Ages and Stages Questionnaire-Social Emotional (ASQ-SE-2) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The ASQ-SE-2 is a 26-item, parent-completed questionnaire that is highly reliable and focuses solely on social-emotional development in young children aged 1-72 months.
Children's developmental functioning will be measured using the Ages and Stages Questionnaire-Third Edition (ASQ-3) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The ASQ-3 consists of a series of parent-completed questionnaires to assess child development across ﬁve domains for children 1 to 66 months: communication, gross motor, ﬁne motor, problem-solving, and personal-social skills.

SECONDARY OUTCOMES:
Children's exposure to risk and protective factors will be measured using a cumulative risk measure (Bondi et al., 2020) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  This cumulative risk measure is designed to identify risk and protective factors for children of substance-involved mothers. It will be used to assess children's exposure to risk (e.g., ACEs, poverty, maternal mental illness) and protective factors (e.g., family social support, childcare, community supports).
Sensitivity of maternal behaviour will be measured using the Maternal Behavior Q-Sort (MBQS) Brief Version | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The MBQS Brief Version is composed of 25 items and will be used by researchers to assess the sensitivity of maternal behaviour from a 10-minute in vivo mother-child interaction.
Maternal stress will be measured using the Parenting Stress Index Short Form (PSI-4-SF) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The PSI-4-SF consists of 36 items. All domains (Parent Distress, Difﬁcult Child, and Parent-Child Dysfunctional Interaction) and the Total Stress Scale have acceptable reliability and validity.
Parenting attitudes will be measured using the Adult-Adolescent Parenting Inventory Version 2.0 (AAPI-2) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The AAPI-2 is composed of 40 items and will be used to assess parenting attitudes related to expectations, empathy, and discipline.
Self-efficacy and satisfaction as a parent will be measured using the Being a Parent Scale | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The Being a Parent Scale consists of 16 items.
Quality and quantity of stimulation available to the child will be measured using the Home Observation for Measurement of the Environment Inventory (HOME) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The HOME is a 45-item questionnaire designed to measure the quality and quantity of stimulation available to young children.
Maternal depression will be measured using the Center for Epidemiological Studies Depression Scale (CES-D) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The CES-D consists of 20 items.
Maternal anxiety will be measured using the Beck Anxiety Inventory (BAI) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The BAI consists of 21 items.
Maternal adverse childhood experiences (ACEs) will be measured using a Maternal ACEs Measure (Felitti et al., 1998; Dube et al., 2003) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  This 10-item questionnaire requires mothers to retrospectively report on their ACEs prior to 18 years of age. The questions pertain to abuse, neglect, and household dysfunction.
Maternal anxiety will be measured using the Generalized Anxiety Disorder Scale (GAD-7) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The GAD-7 consists of 7 items.
Maternal depression will be measured using the Patient Health Questionnaire-9 (PHQ-9) | Change from pre-intervention to 12 months after engagement and 24 months after engagement
  The PHQ-9 consists of 9 items.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Maxxine Wright Community Health Centre, Surrey, British Columbia
  - Mothercraft, Breaking the Cycle, Toronto, Ontario

REFERENCES:
- [Derived] Racine N, Barriault S, Motz M, Leslie M, Poole N, Premji S, Andrews NCZ, Penaloza D, Pepler D. A comparative effectiveness study of the breaking the cycle and Maxxine Wright intervention programs for substance-involved mothers and their children: study protocol. BMC Psychol. 2024 Jan 5;12(1):16. doi: 10.1186/s40359-023-01484-w. PMID 38183089